CLINICAL TRIAL: NCT05026203
Title: Effectiveness of Ketamine Treatment in Difficult-to-treat Depression Comparing With Midazolam: a Double-blind Randomized Controlled Trial and Its Cost Effectiveness Analysis
Brief Title: Effectiveness of Ketamine Treatment for Three Consecutive Days in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Keerati Pattanaseri, Consualtant psychiatrist, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109/2564(IRB1)
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental)
  Interventions: Drug: Ketamine Hydrochloride
- Midazolam (Placebo Comparator)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Ketamine hydrochloride 0.5 mg/kg intravenous administer in 40 minutes per day for 3 consecutive days
  Arms: Ketamine
Drug: Midazolam — Midazolam
  Arms: Midazolam

SUMMARY:
Inclusion criteria: 1. patient over 20 years old with depression diagnosed by a psychiatrist and MADRS >= 25 scores; 2. failed to improve by at least optimal dosage of two antidepressants for four weeks and one psychotherapy. Patients and outcome assessors will be blinded from intervention the patients have.

Participants will be randomized into two groups that are intervention (ketamine 0.5 mg/kg IV drip in 40 minutes) and control (midazolam 0.045 mg/kg IV drip in 40 minutes) groups. Participants will administer ketamine/midazolam once daily for three consecutive days. They will be evaluate MADRS changing, vital signs, dissociative symptoms, CGI, and quality of life (EQ-5D-5L) during the treatment, at 1 week and 4 weeks after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* over 20 years old
* depression was diagnosed by a psychiatrist and having MADRS >= 25
* depression treated with 2 optimal dosage of antidepressants for 4 weeks and one psychotherapy
* stable dosage of current medications for 4 weeks
* fluently Thai

Exclusion Criteria:

* secondary depression
* PTSD
* current pregnancy
* history of increased intracranial hemorrhage, increased intracranial pressure, severe head injury, abnormal thyroid function, angina, heart failure, arrhythmia, aneurysm, uncontrolled hypertension, chronic lower tract respiratory disease, myasthenia gravis, glaucoma, dementia, acute porphyria, or cystitic (within 3 months prior to recruitment)
* allergy to ketamine or midazolam
* history of substance use disorder within 1 year prior to recruitment
* history of psychosis within 3 months
* history of bipolar disorder
* BMI over 35
* frail medical condition
* currently ECT or TMS

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | 1 month
  decrease more than 50% of scale from baseline is defined as remission

SECONDARY OUTCOMES:
dissociation | immediately after administraion
  The dissociative experiences measure, Oxford (DEMO)
health questionnaire | 1 month
  The 5-level EQ-5D version (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Locations (1):
- Keerati Pattanaseri, Bangkok, Thailand

REFERENCES:
- [Derived] Pattanaseri K, Lortrakul J, Jaisin K, Srifuengfung M, Sa-Nguanpanich N, Viravan N, Pariwatcharakul P, Makarasara W, Ratta-Apha W. A randomized controlled pilot study of daily intravenous ketamine over three days for treatment-resistant depression. BMC Psychiatry. 2024 Jul 18;24(1):512. doi: 10.1186/s12888-024-05951-5. PMID 39026266